CLINICAL TRIAL: NCT06617845
Title: Optimizing Brain Stimulation Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian N. Lundstrom, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-009654
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stimulation set A/B group (Experimental): Device will be set to use stimulation parameters from set A first (e.g. 145 Hz) and then from set B (e.g. low frequency stimulation).
  Interventions: Device: Stimulation Set A and B
- Stimulation set B/A group (Experimental): Device will be set to use stimulation parameters from set B first (e.g. low frequency stimulation) and then from set A (e.g. 145 Hz).
  Interventions: Device: Stimulation Set A and B

INTERVENTIONS:
Device: Stimulation Set A and B — Subjects will receive one stimulation parameter set first for 3 months and then the other for three months. Sets will include Set A (145 Hz high frequency stimulation) and Set B (Low frequency stimulation less than 40 Hz, which is similar to stimulation frequencies used during cortical stimulation). The 145 Hz stimulation will be set to cycling (1 min on, 5 min off) while the low frequency setting will be continuous. Both sets include stimulation parameter sets that have been used in clinical practice as a part of standard of care. However, it is unclear which set is better or whether they are similarly effective.

SUMMARY:
A primary purpose of this study is to better understand what stimulation parameters work best for patients. For example, for Deep Brain Stimulation (DBS) of the Anterior Nucleus of the Thalamus (ANT), it is not clear what stimulation frequency leads is most effective. This study will help assess the effectiveness of low frequency or high frequency stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are implanted with a brain stimulation device targeting the anterior nucleus of the thalamus per Mayo Clinic standard of care

Exclusion Criteria:

* Patients for whom clinical follow-up is not expected during the initial 6-8 months following implant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Seizure burden | Baseline, 4 months, 7 months, 12 months
  Using the Mayo Epilepsy Short Assessment as well as patient diaries, seizure frequency is determined.

SECONDARY OUTCOMES:
Change in Mayo Post-Stimulation Activation score | Baseline, 4 months, 7 months, 12 months
  The Mayo Post-Stimulation Activation questionnaire is a 9-item survey measuring post-stimulation symptoms such as speech problems, numbness, muscle tightness, balance, lightheadedness, vision, mood changes, and memory. The questionnaire is ranked on a Likert scale of 1 - Mild; 2 - Moderate; 3 - Severe; 4 - N/A. The minimum value is 1 and the maximum value is 4, where 1 represents less severe.
Change in Mayo Epilepsy Short Assessment (MESA) score | Baseline, 4 months, 7 months, 12 months
  The Mayo Epilepsy Short Assessment (MESA) is a questionnaire measuring seizure frequency, seizure severity, quality of life, sleep, and mood. Seizure frequency is measured by number of seizures per month. Severity, life satisfaction, and sleep quality are measured from 1 (worst) to 10 (best). Mood and anxiety are measured on a 4-point scale with the following options (Not at all, Several days, More than half the days, Nearly every day).

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Optimizing stimulation parameters for anterior thalamic nuclei deep brain stimulation in epilepsy: A randomized crossover trial — http://pubmed.ncbi.nlm.nih.gov/40423665/